CLINICAL TRIAL: NCT00630682
Title: A Pilot Trial of Dextroamphetamine for Methamphetamine Dependence
Acronym: 1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Gantt Galloway, PharmD, Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25.139; P50DA018179 (NIH)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Methamphetamine Addiction
Keywords: Methamphetamine; Drug Abuse; Drug Treatment; Addiction; Meth; Treatment for Methamphetamine Dependence
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextroamphetamine (Active Comparator): Active drug
  Interventions: Drug: Dextroamphetamine
- Placebo (Placebo Comparator): Placebo of drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextroamphetamine — 1 week placebo and 8 weeks 60mg d-AMP QD.
  Arms: Dextroamphetamine
Drug: Placebo — 9 weeks of placebo 60mg capsules QD.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness dextroamphetamine to help methamphetamine users quit or cut down on their use. The study lasts for 9 weeks. Eligible participants will attend research visits twice per week, and will receive individual counseling sessions once per week for all 9 weeks. 50% of the participants will receive the active medication while the other 50% will receive the placebo (sugar pill). Neither the participant or the study team will know if the participant is receiving the placebo or active drug.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 yrs. old

Exclusion Criteria:

* pregnant or lactating females

  * Contact site for additional information

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Subjects treated with dextroamphetamine will have better outcomes than subjects treated with placebo, as indicated by the number of urine samples that do not indicate new use of MA (the primary outcome measure) | Twice per week for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gantt Galloway, PharmD, Principal Investigator — Addiction Pharmacology Research Laboratory
Locations (1):
- CPMC-St. Luke's Campus-Addiction Pharmacology Research Laboratory, San Francisco, California, United States